CLINICAL TRIAL: NCT00463229
Title: The Comparative Acceptability, Safety, Effects and Expense of Specialized, Integrated, and Interdisciplinary Community Rehabilitation for Stroke Survivors and Their Caregivers
Brief Title: Interdisciplinary Team Approach to Stroke Rehabilitation in Home Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Ministry of Health and Long Term Care (Other Government); Toronto Central Community Care Access Centre (Other); Heart and Stroke Foundation of Ontario (Other); Greater Toronto Area Rehabilitation Network (Unknown)
Responsible Party: Principal Investigator, Maureen Markle-Reid, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHE-78692
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; home care services; effectiveness; quantitative research; interdisciplinary; cost; health services research, integrated
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interprofessional Team Approach (Experimental): Participants in the experimental group will receive home care services from a team of professional service providers [Community Care Access Centre (CCAC) Care Coordinator, Registered Nurse, Occupational therapist, Physiotherapist, Speech language pathologist, Nutritionist] and non-professional service providers (personal support workers) with experience and training in stroke care. The team will provide a comprehensive, coordinated and evidence-based approach to stroke rehabilitation through weekly case conferencing, a written interdisciplinary care plan, and joint visits.
  Interventions: Other: Interprofessional Team Approach
- Usual Home Care Services (No Intervention): Participants allocated to the control group received standard home care services arranged by the CCAC. These include routine follow-up by the CCAC case manager whose focus is on assessment and referral to community agencies, and ongoing monitoring and evaluating the plan of care through in-home assessment with clients.

INTERVENTIONS:
Other: Interprofessional Team Approach — Subject in the second group will receive home care services from a team of professional service providers (CCAC Care Coordinator, Registered Nurse, Occupational therapist, Physiotherapist, Speech language pathologist, Nutritionist) and non-professional service providers (personal support workers) with experience and training in stroke care. The team will provide a comprehensive, coordinated and evidence-based approach to stroke rehabilitation through weekly case conferencing, a written interdisciplinary care plan, and joint visits.
  Other Names: Interdisciplinary Stroke Rehabilitation Team
  Arms: Interprofessional Team Approach

SUMMARY:
As the population ages and the number of stroke survivors increases, information is needed to determine the best way of providing home care services for rehabilitation to stroke survivors and their caregivers while containing health care costs. This project will address this area by developing and testing the effects and costs of a collaborative and specialized team approach to stroke rehabilitation by health professionals, in a home care setting, compared to usual home care services. The overall goal of this way of providing home care services is to improve the quality of life and function of stroke survivors and their caregivers and prevent future strokes, which will reduce the overall cost to the health care system.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death in Canada, and is considered to be the most common disabling chronic condition. Approximately 40,000 to 50,000 people in Canada experience a stroke each year and about 80% of these people survive. Many of these people who survive a stroke never fully recover and are left with significant impairments and disabilities, and 12% to 25% will have another stroke within the first year. This results in a significant burden to individuals, families, and society as a whole. Of every 100 people who are hospitalized for a stroke, 15-40 return home and require home care services for rehabilitation. Stroke rehabilitation is one of the key components of stroke care. The goal of rehabilitation is to assist stroke survivors to reach his or her optimal level of physical, social, and emotional function.

Information gained from this study will be used to inform home care practice, policy decisions and the allocation of home care resources and make a national contribution to health care delivery reform.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke or TIA has been confirmed.
* newly referred to and eligible for home care services (physiotherapy, speech language therapy, occupational therapy, nursing) through the Toronto Central CCAC.
* living at home in the community (outside of an institutional setting) up to 18-months post-stroke.
* English speaking

Exclusion Criteria:

* refuse to give informed consent.
* more than 18 months post-stroke at time of recruitment.
* unable to read/write English and an appropriate translator is not available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Markle-Reid, RN MScN PhD, Principal Investigator — McMaster University, School of Nursing
Locations (1):
- School of Nursing, McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Markle-Reid M, Orridge C, Weir R, Browne G, Gafni A, Lewis M, Walsh M, Levy C, Daub S, Brien H, Roberts J, Thabane L. Interprofessional stroke rehabilitation for stroke survivors using home care. Can J Neurol Sci. 2011 Mar;38(2):317-34. doi: 10.1017/s0317167100011537. PMID 21320840

RESULTS

PARTICIPANT FLOW:
Groups:
- Interprofessional Team Approach: Participants in the experimental group will receive home care services from a team of professional service providers (CCAC Care Coordinator, Registered Nurse, Occupational therapist, Physiotherapist, Speech language pathologist, Nutritionist) and non-professional service providers (personal support workers) with experience and training in stroke care. The team will provide a comprehensive, coordinated and evidence-based approach to stroke rehabilitation through weekly case conferencing, a written interdisciplinary care plan, and joint visits.
Period: Overall Study
Arm/Group | Interprofessional Team Approach | Usual Home Care Services
Started | 52 | 49
Completed | 43 | 39
Not Completed | 9 | 10
Not completed — Lost to Follow-up | 5 | 7
Not completed — Death | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interprofessional Team Approach | Usual Home Care Services | Total
Number analyzed (Participants) | 52 | 49 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 23
  >=65 years | 42 | 36 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.18 (12.35) | 72.32 (14.14) | 74.31 (13.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 27 | 27 | 54
Region of Enrollment [Number; unit: participants]
  Canada | 52 | 49 | 101

OUTCOME MEASURES:

1. Primary Outcome: Change Between the Value of the SF-36 Physical Function Score at 12 Months Minus Value at Baseline to Measure the Change in Health-related Quality of Life and Function
Description: The primary measure of effect was the change in health-related quality of life and functioning from baseline to 12-months as measured by the SF-36 physical functioning score. The range of possible scores for this subscale is 0-100, with a higher score indicating a more favourable health status.
Time Frame: Baseline (pre-randomization) and 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Interprofessional Team Approach | Usual Home Care Services
Number analyzed (Participants) | 43 | 39
Units on a scale | 28.84 (30.68) | 28.85 (28.48)

2. Secondary Outcome: Stroke Impact Scale - 16
Description: The SIS-16 assesses several aspects of health-related quality of life that are important to stroke survivors, caregivers, and healthcare professionals. The SIS-16 consists of 16 items which cover the physical aspects of stroke including: strength, hand function, mobility, and activities of daily living/instrumental activities of daily living. Each item is assigned a score ranging from 1 (could not do at all) to 5 (not difficult at all). The individual items sum to provide a total score (range from 16 to 80), with higher scores indicating higher levels of health-related quality of life and function.
Time Frame: Baseline (pre-randomization) and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interprofessional Team Approach | Usual Home Care Services
Number analyzed (Participants) | 43 | 39
units on a scale | -2.11 (16.65) | -0.49 (18.81)

3. Secondary Outcome: Reintegration to Normal Living Index
Description: The RNLI assesses global functional status and measures both the stroke survivors' perceptions of their own capabilities and objective indicators of physical, social, and psychological performance. The RNLI consists of 11 items which cover the domains of mobility, self-care abilities, daily activities, recreational and social activities, family roles, and personal relationships, presentation of self and general coping skills. Each item is scored as 0 to 2. Minimum score is "0" and maximum score is "22". The individual items sum to provide a total score, with 22 indicating the highest degree of reintegration.
Time Frame: Baseline (pre-randomization) and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interprofessional Team Approach | Usual Home Care Services
Number analyzed (Participants) | 43 | 39
units on a scale | 14.84 (5.71) | 15.44 (5.29)

4. Secondary Outcome: Short Portable Mental Status Questionnaire.
Description: The 10-item Short Portable Mental Status Questionnaire (SPMSQ) is used for the screening, diagnosis and assessment of cognition. The SPMSQ is short, easily administered and has been designed, tested, standardized and validated in a variety of populations, including stroke. The SPMSQ consists of 10 items. The individual items sum to provide a total score, ranging from 0-10; with greater than 4 errors indicating some degree of intellectual impairment. The higher the score, the less impairment.
Time Frame: Baseline (pre-randomization) and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interprofessional Team Approach | Usual Home Care Services
Number analyzed (Participants) | 43 | 39
units on a scale | 0.38 (2.17) | 0.67 (1.38)

5. Secondary Outcome: Centre for Epidemiological Studies in Depression Scale (CES-D)
Description: The CES-D scale is a 20-item, self-reported questionnaire that assesses the current frequency of depressive symptoms. Total scores can range from 0 to 60; the higher the score, the more depressed. Values were determined by taking the value of the 12-month data (Timepoint 2) and subtracting them from the baseline data (Timepoint 1).
Time Frame: Baseline and 12 months
Population: Timepoint 2 minus Timepoint 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interprofessional Team Approach | Usual Home Care Services
Number analyzed (Participants) | 43 | 39
units on a scale | -2.77 (9.52) | -2.13 (9.34)

6. Secondary Outcome: Personal Resource Questionnaire (PRQ85-Part Two)
Description: The PRQ85-Part Two is a 25-item scale that measures perceived social support along five dimensions: provision for attachment/intimacy; social integration; opportunity for nurturing behaviour; reassurance of worth as an individual and in role accomplishments; and the availability of informational, emotional, and material help. Scores range from a minimum of 25 to maximum score of 175; a higher score indicates a greater perception of social support.
Time Frame: Baseline (pre-randomization) and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interprofessional Team Approach | Usual Home Care Services
Number analyzed (Participants) | 43 | 39
units on a scale | 4.5 (14.09) | 1.01 (17.74)

7. Secondary Outcome: Kessler - 10
Description: The Kessler-10 assesses level of anxiety and depressive symptoms a person may have experienced in the most recent four-week period. Its main strength is a superior ability to screen for anxiety and affective disorders. Each item is assigned a score ranging from 5 (all of the time) to 1 (none of the time). These 10 items are summed to give scores ranging from 10-50, where 50 indicates high risk of anxiety or depressive disorder. Previous studies have established a cut-off score of 16-29/50 for medium risk, and 30-50/50 as high risk for anxiety and depressive disorders.
Time Frame: Baseline (pre-randomization) and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interprofessional Team Approach | Usual Home Care Services
Number analyzed (Participants) | 43 | 39
units on a scale | -1.66 (4.79) | -0.46 (5.3)

ADVERSE EVENTS:
Arm/Group | Interprofessional Team Approach | Usual Home Care Services
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49
Other Adverse Events (participants affected / at risk) | 0/52 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes